CLINICAL TRIAL: NCT05528081
Title: A Longitudinal Follow-up Study of the Patients With Medication-overuse Headache or Migraine That Completed Baseline MRI
Brief Title: Longitudinal Study of the Patients With Medication-overuse Headache or Migraine That Completed Baseline MRI
Acronym: LMMM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wei Dai (Other)
Collaborators: International Headache Society (Unknown)
Responsible Party: Sponsor-Investigator, Wei Dai, Principal Investigator Wei Dai, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: S-2022-543-01
Record Dates: First submitted 2022-08-20; First posted 2022-09-06 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Migraine Disorders; Medication-overuse Headache
Keywords: Migraine; Medication-overuse Headache; MRI
MeSH Terms: conditions — Migraine Disorders; Headache Disorders, Secondary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Persons with migraine disease: Persons diagnosed with migraine based on the third edition of the International Classification of Headache Disorders (ICHD-3) and underwent baseline 3-tesla MRI
  Interventions: Other: Phone interview
- Persons with medication-overuse headache: Persons diagnosed with MOH based on the ICHD-3 and underwent baseline 3-tesla MRI
  Interventions: Other: Phone interview
- Healthy controls: Healthy individuals with no history of primary or secondary headache based on the ICHD-3 and underwent baseline 3-tesla MRI

INTERVENTIONS:
Other: Phone interview — Participants will be interviewed by phone at 3, 12, 24 months after the baseline MRI scans.
  Groups: Persons with medication-overuse headache; Persons with migraine disease

SUMMARY:
This is a phone interview research study for patients with migraine or medication-overuse headache (MOH) who have completed baseline MRI scans. Participants will be interviewed by phone at 3, 12, 24 months after the baseline MRI scans.

The purpose of this study is to potentially identify the baseline brain functional or structural signatures (functional connectivity, regional homogeneity, amplitude of low frequency fluctuation, and so such) that are predictive of the short- and long- term outcomes as well as treatment response of migraine and MOH patients.

DETAILED DESCRIPTION:
Participants have been administered informed consent, taken medical history and performed a physical examination, and completed MRI scans at baseline visit. This study only comprises the follow-up research procedure.

After the MRI scans, all included patients were treated at the headache center by headache specialists according to their clinical experience. The follow-up time points will be 3 months, 12 months, 24 months after baseline MRI scans. The investigator will interview the patients by telephone to assess their headache features (duration, frequency, severity, accompany symptoms, migraine days per months, moderate to severe headache days per month, medications being used…) and Patient Health Questionnaire 9 Depression Scale (PHQ-9), Generalized Anxiety Disorder Assessment 7-item Scale (GAD-7), quality and patterns of sleep using Pittsburgh Sleep Quality Index (PSQI), and functional disability caused by migraine using the Migraine Disability Assessment Scale (MIDAS) within the last 10 days at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with migraine or MOH at baseline visit, signed the consent form, and completed MRI scans.
* Participants who are willing to take the phone interview during follow-up.

Exclusion Criteria:

* Refuse or unable to complete the phone interview procedure during follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with migraine disease, MOH, and healthy controls who have completed baseline MRI.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Monthly Number of Migraine Days | 3 months after the baseline MRI
  A migraine day is defined as a day with headache lasting at least 30 minutes without intake of analgesics and meeting ICHD-3 criteria for migraine or probable migraine. A migraine day may also be defined as a day with headache that successfully responds to acute treatment with a migraine-specific medication (triptan, ditan, gepant, ergotamine, etc.).
Monthly Number of Migraine Days | 12 months after the baseline MRI
  A migraine day is defined as a day with headache lasting at least 30 minutes without intake of analgesics and meeting ICHD-3 criteria for migraine or probable migraine. A migraine day may also be defined as a day with headache that successfully responds to acute treatment with a migraine-specific medication (triptan, ditan, gepant, ergotamine, etc.).
Monthly Number of Migraine Days | 24 months after the baseline MRI
  A migraine day is defined as a day with headache lasting at least 30 minutes without intake of analgesics and meeting ICHD-3 criteria for migraine or probable migraine. A migraine day may also be defined as a day with headache that successfully responds to acute treatment with a migraine-specific medication (triptan, ditan, gepant, ergotamine, etc.).
Monthly Number of Moderate/Severe Headache Days | 3 months after the baseline MRI
  A moderate/severe headache day is defined as a day with headache pain of moderate or severe intensity that lasts at least 4 hours without medication, or a day with a headache pain of at least moderate intensity that responds to acute treatment with a migraine-specific medication.
Monthly Number of Moderate/Severe Headache Days | 12 months after the baseline MRI
  A moderate/severe headache day is defined as a day with headache pain of moderate or severe intensity that lasts at least 4 hours without medication, or a day with a headache pain of at least moderate intensity that responds to acute treatment with a migraine-specific medication.
Monthly Number of Moderate/Severe Headache Days | 24 months after the baseline MRI
  A moderate/severe headache day is defined as a day with headache pain of moderate or severe intensity that lasts at least 4 hours without medication, or a day with a headache pain of at least moderate intensity that responds to acute treatment with a migraine-specific medication.
Severity of Headache Measured by Visual Analogue Scale | 3 months after the baseline MRI
  Severity of headache is measured by VAS ranging from 0 to 10 with 1 = most mild to 10 = most severe. The mean severity of headache for each month will be calculated as: sum of severity of headache days divided by number of headache days.
Severity of Headache Measured by Visual Analogue Scale | 12 months after the baseline MRI
  Severity of headache is measured by VAS ranging from 0 to 10 with 1 = most mild to 10 = most severe. The mean severity of headache for each month will be calculated as: sum of severity of headache days divided by number of headache days.
Severity of Headache Measured by Visual Analogue Scale | 24 months after the baseline MRI
  Severity of headache is measured by VAS ranging from 0 to 10 with 1 = most mild to 10 = most severe. The mean severity of headache for each month will be calculated as: sum of severity of headache days divided by number of headache days.
Mean Headache Duration (hours) | 3 months after the baseline MRI
  As a feature of the headache attack duration.
Mean Headache Duration (hours) | 12 months after the baseline MRI
  As a feature of the headache attack duration.
Mean Headache Duration (hours) | 24 months after the baseline MRI
  As a feature of the headache attack duration.
Nausea (number) | 3 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Nausea (number) | 12 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Nausea (number) | 24 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Vomiting (number) | 3 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Vomiting (number) | 12 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Vomiting (number) | 24 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Photophobia (number) | 3 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Photophobia (number) | 12 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Photophobia (number) | 24 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Phonophobia (number) | 3 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Phonophobia (number) | 12 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Phonophobia (number) | 24 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Aggravation by Movement (number) | 3 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Aggravation by Movement (number) | 12 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Aggravation by Movement (number) | 24 months after the baseline MRI
  As a feature of the accompany symptoms during an attack.
Response to Acute Treatment | 3 months after the baseline MRI
  To describe response to prior acute medications.
Response to Acute Treatment | 12 months after the baseline MRI
  To describe response to prior acute medications.
Response to Acute Treatment | 24 months after the baseline MRI
  To describe response to prior acute medications.
Response to Prophylactic Treatment | 3 months after the baseline MRI
  To describe response to prior prophylactic medications.
Response to Prophylactic Treatment | 12 months after the baseline MRI
  To describe response to prior prophylactic medications.
Response to Prophylactic Treatment | 24 months after the baseline MRI
  To describe response to prior prophylactic medications.
Migraine Disability Assessment Test Total Score | 3 months after the baseline MRI
  The MIDAS was designed to quantify headache-related disability over a 3-month period. This instrument consists of 5 items that measures the impact that migraine headaches have on patients' life, including days of work/school missed, days with productivity at work/school reduced to half or more, days with household work missed, days with productivity in household work reduced to half or more, and days missed family/social/leisure activities. Each item has a numeric response range from 0 to 90 days; if days are missed from work/school or household work they are not counted as days with reduced productivity at work/school or household work. The numeric responses are summed to produce a total score ranging from 0 to 270. A higher value is indicative of more disability.
Migraine Disability Assessment Test Total Score | 12 months after the baseline MRI
  The MIDAS was designed to quantify headache-related disability over a 3-month period. This instrument consists of 5 items that measures the impact that migraine headaches have on patients' life, including days of work/school missed, days with productivity at work/school reduced to half or more, days with household work missed, days with productivity in household work reduced to half or more, and days missed family/social/leisure activities. Each item has a numeric response range from 0 to 90 days; if days are missed from work/school or household work they are not counted as days with reduced productivity at work/school or household work. The numeric responses are summed to produce a total score ranging from 0 to 270. A higher value is indicative of more disability.
Migraine Disability Assessment Test Total Score | 24 months after the baseline MRI
  The MIDAS was designed to quantify headache-related disability over a 3-month period. This instrument consists of 5 items that measures the impact that migraine headaches have on patients' life, including days of work/school missed, days with productivity at work/school reduced to half or more, days with household work missed, days with productivity in household work reduced to half or more, and days missed family/social/leisure activities. Each item has a numeric response range from 0 to 90 days; if days are missed from work/school or household work they are not counted as days with reduced productivity at work/school or household work. The numeric responses are summed to produce a total score ranging from 0 to 270. A higher value is indicative of more disability.
Patient Health Questionnaire 9 Depression Scale Total Score | 3 months after the baseline MRI
  The PHQ-9 was designed to identify signs or symptoms of depression over a two-week period. The total score is calculated and can range from zero to 27. Scores of 5, 10, 15, and 20 are taken as the cut-off points for mild, moderate, moderate to severe, and severe depression, respectively.
Patient Health Questionnaire 9 Depression Scale Total Score | 12 months after the baseline MRI
  The PHQ-9 was designed to identify signs or symptoms of depression over a two-week period. The total score is calculated and can range from zero to 27. Scores of 5, 10, 15, and 20 are taken as the cut-off points for mild, moderate, moderate to severe, and severe depression, respectively.
Patient Health Questionnaire 9 Depression Scale Total Score | 24 months after the baseline MRI
  The PHQ-9 was designed to identify signs or symptoms of depression over a two-week period. The total score is calculated and can range from zero to 27. Scores of 5, 10, 15, and 20 are taken as the cut-off points for mild, moderate, moderate to severe, and severe depression, respectively.
Generalized Anxiety Disorder Assessment 7-item Scale Total Score | 3 months after the baseline MRI
  The GAD-7 was designed to identify signs or symptoms of anxiety over a two-week period. The total score is calculated and can range from zero to 21. Scores of 5, 10, 14, and 19 are taken as the cut-off points for mild, moderate, moderate to severe, and severe anxiety, respectively.
Generalized Anxiety Disorder Assessment 7-item Scale Total Score | 12 months after the baseline MRI
  The GAD-7 was designed to identify signs or symptoms of anxiety over a two-week period. The total score is calculated and can range from zero to 21. Scores of 5, 10, 14, and 19 are taken as the cut-off points for mild, moderate, moderate to severe, and severe anxiety, respectively.
Generalized Anxiety Disorder Assessment 7-item Scale Total Score | 24 months after the baseline MRI
  The GAD-7 was designed to identify signs or symptoms of anxiety over a two-week period. The total score is calculated and can range from zero to 21. Scores of 5, 10, 14, and 19 are taken as the cut-off points for mild, moderate, moderate to severe, and severe anxiety, respectively.
Quality and Patterns of Sleep Using Pittsburgh Sleep Quality Index Total Score | 3 months after the baseline MRI
  The PSQI is to assess sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for the seven components yields one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Quality and Patterns of Sleep Using Pittsburgh Sleep Quality Index Total Score | 12 months after the baseline MRI
  The PSQI is to assess sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for the seven components yields one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Quality and Patterns of Sleep Using Pittsburgh Sleep Quality Index Total Score | 24 months after the baseline MRI
  The PSQI is to assess sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for the seven components yields one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Dai, M.D., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided